CLINICAL TRIAL: NCT04571359
Title: Relationship of Spot Urine Oxalate to Creatinine Ratio and 24 Hours Urinary Oxalate Excretion in Patients With Urolithiasis
Brief Title: Spot Urine Oxalate to Creatinine Ratio and 24 Hours Urinary Oxalate
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Syed bilal hashmi, Resident, Aga Khan University
Other Study IDs: 5084-Pat-ERC-17
Record Dates: First submitted 2020-09-27; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Urolithiasis; Hyperoxaluria
Keywords: 24-hour urinary oxalate; Spot oxalate to creatinine ratio
MeSH Terms: conditions — Urolithiasis; Hyperoxaluria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Oxalate to creatinine ratio — Comparsion between 24 hours urine oxalate and spot urine oxalate to creatinine ratio

SUMMARY:
The evaluation of 24 hour urinary oxalate excretion is the gold standard for diagnosing Hyperoxaluria in patients with recurrent urolithiasis. The relationship of oxalate measurement between spot and 24 hour urine sample has not been studied in Pakistani population before. Thus, it is necessary to see if spot urine samples show good correlation with 24 hour urine samples in our population where the frequency of hyperoxaluria in patients with urolithiasis is reported to be 64.5%. Also, the various pre analytical issues associated with 24 hour urinary collection which may lead to the incorrect or misdiagnosis, need for duplicate testing consuming extra resources and man power. We therefore, in this study, want to see the correlation between 24 hour urinary oxalate and oxalate to creatinine ratio. The aim of our study is to determine the relationship between 24 hour urinary oxalate and spot urine oxalate to creatinine ratio and to identify if oxalate to creatinine ratio can be used as an alternative to 24 hour urinary oxalate

DETAILED DESCRIPTION:
A cross-sectional study was conducted at Section of Chemical Pathology, Department of Pathology and Laboratory Medicine, Aga Khan University, Karachi from 1st February to 31st December 2019. Adult patients with history of kidney stones presenting at the Clinical Laboratory for 24 hours urine oxalate estimation were included in the study. Debilitated or bed ridden patients and patients with renal failure or end stage renal disease, in whom urinary oxalate is no longer an indicator of disease status were excluded from the study. Study was approved by ethical review committee of Aga Khan University Hospital. Patients after informed consent, were guided to submit a spot urine sample. Clinical details were recorded on a structured questionnaire by the principal investigator.

24 hour urine samples were collected in a jar having thymol, which is routinely added to limit bacterial growth and hence guard against citrate degradation. Spot urine samples were collected in red top container without any added preservatives. The specimen were transported to the laboratory within the 12 hours of collection of 24 hour urinary specimen.

Volume of 24 hour urine was measured in liters. After mixing of the urinary sample to overcome effects of sedimentation, a 6 ml aliquot was made and HCl was added to avoid the precipitation of oxalate crystals in every sample. Specimen was stored at -20 C till further analysis.

Urinary oxalate was measured on Micro lab 300 using a kit based on oxalate oxidase principle by Trinity Biotech plc. Wick low, Ireland following standard operating procedures. Urinary creatinine was measured on ADVIA 1800 by Siemens, US using kinetic Jaffe reaction. Both normal and abnormal quality control materials were run with every batch of oxalate and creatinine analysis in urine to validate the results. In addition, external proficiency testing of urinary oxalate was conducted by College of American Pathologists (CAP).

The cut-offs for 24 hour oxalate excretion was 502 ųmol/24 hours for males and 353 ųmol/24 hours for females. The cut-offs for spot oxalate: creatinine ratio was 33 ųmol/mmol for males and 45 ųmol/mmol for females.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of kidney stones.
* All patients investigated for 24 hour urinary oxalate excretion.
* Patients between 18 years to 60 years would be included.
* Both genders will be included.

Exclusion Criteria:

* Debilitated patients or bed ridden patients in whom proper and complete 24 hour urine collection will be troublesome.
* Patients with renal failure/end stage renal disease, in whom urinary oxalate is no longer an indicator of disease status.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients with history of kidney stones presenting at the Clinical Laboratory for 24 hours urine oxalate estimation.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Relationship between 24 hour urinary oxalate excretion and spot urine oxalate to creatinine ratio | 1 year
  Relationship between 24 hour urinary oxalate excretion and spot urine oxalate to creatinine ratio to determine its clinical utility against the use of 24 hour urinary oxalate estimation which is the standard practice.

CONTACTS AND LOCATIONS:
Overall Officials: Syed bilal hashmi, Principal Investigator — AKUH
Locations (1):
- Syed bilal hashmi, Karachi, Pakistan, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hagler L, Herman RH. Oxalate metabolism. I. Am J Clin Nutr. 1973 Jul;26(7):758-65. doi: 10.1093/ajcn/26.6.758. No abstract available. PMID 4576881
- [Background] Hoppe B. An update on primary hyperoxaluria. Nat Rev Nephrol. 2012 Jun 12;8(8):467-75. doi: 10.1038/nrneph.2012.113. PMID 22688746